CLINICAL TRIAL: NCT02683187
Title: Role of Alpha-cell GLP-1 in the Beta-cell Response to DPP-4 Inhibition
Brief Title: DPP4 Inhibition & Beta Cell Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David D'Alessio, M.D. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, David D'Alessio, M.D., Professor, Division Chief of Endocrinology Division, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00067061
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: insulin secretion; GLP-1; alpha cell; paracrine effect; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Active Comparator): The infusion procedures performed during study visits 2 and 3 are identical except that the oral medicine Sitagliptin will only be administered at one of the two visits, with order of Sitagliptin administration determined at random by study staff. In this arm, Sitagliptin will be administered.
  Interventions: Drug: Active Comparator: Sitagliptin
- Non-Sitagliptin (Placebo Comparator): The infusion procedures performed during study visits 2 and 3 are identical except that the oral medicine Sitagliptin will only be administered at one of the two visits, with order of Sitagliptin administration determined at random by study staff. In this arm, placebo will be administered
  Interventions: Drug: Placebo Comparator - No Sitagliptin

INTERVENTIONS:
Drug: Active Comparator: Sitagliptin — Subjects will receive sitagliptin prior to the start of the experiment involving 1/2 of the subjects receiving Exendin-9 (a GLP-1 receptor blocker) first over 60 minutes ; followed by a bolus arginine (5g) infusion after 30 minutes into the Ex-9 infusion, with blood draws over the next 30 minutes. Followed by a 60 minute washout and the procedure is repeated , this time with saline instead of Ex-9 (these procedures are reversed - saline first then Ex-9 - half of the time).
  Arms: Sitagliptin
Drug: Placebo Comparator - No Sitagliptin — Subjects will receive Placebo (instead of sitagliptin) prior to the start of the experiment involving 1/2 of the subjects receiving Exendin-9 (a GLP-1 receptor blocker) first over 60 minutes ; followed by a bolus arginine (5g) infusion after 30 minutes into the Ex-9 infusion, with blood draws over the next 30 minutes. Followed by a 60 minute washout and the procedure is repeated , this time with saline instead of Ex-9 (these procedures are reversed - saline first then Ex-9 - half of the time).
  Arms: Non-Sitagliptin

SUMMARY:
This study is being done to determine the role of a hormone, glucagon-like peptide 1 (GLP-1), on insulin secretion and to study how GLP-1 works in in diabetic individuals as compared to non-diabetic individuals, under fasting conditions.

GLP-1 is a naturally occurring hormone made in the intestines. It is released into the circulating blood after eating and helps to control the blood glucose levels by increasing insulin secretion by cells in the pancreas. However, the exact method by which GLP-1 causes insulin secretion and how GLP-1 activity is changed in diabetic persons remain unclear. This research is being done to address these questions and better understand the function of GLP-1.

In this research, the investigators will use a synthetic form of Exendin-9 to determine the effects of GLP-1 on insulin secretion in diabetic and non-diabetic persons. Exendin-9 acts as a blocker of GLP-1 action, allowing us to study the specific effects of the GLP-1 hormone. Exendin-9 is an investigational compound, which means it is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA).

In this study, the investigators will also use the drug Sitagliptin, which is an FDA-approved drug for the treatment of type 2 diabetes mellitus. In this study, use of Sitagliptin is considered investigational since it is not being used for treatment of diabetes but is instead being used to understand how GLP-1 works and to better understand how medications like Sitagliptin work in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic cohort: adults age 35-70 years with Type 2 diabetes managed by an oral medication or diet and exercise
* Non-diabetic cohort: healthy adults age 35-70 years
* Male or female
* Ability to speak and understand English
* Diabetic cohort: HbA1c ≤ 8.0%
* Non-diabetic cohort: HbA1c ≤ 6.2%

Exclusion Criteria:

* Rheumatoid arthritis
* Inflammatory bowel disease
* Unstable angina or uncompensated heart failure
* Pulmonary disorders, including COPD and asthma
* Malabsorptive GI disease, such as celiac disease, or gastric bypass
* Significant hepatic disease
* Renal insufficiency (eGFR < 60 mL/kg/min)
* Anemia (hematocrit < 34%) as measured at screening visit
* Uncontrolled hypertension
* Pregnant females
* Consumption of daily medications that alter glucose metabolism of GI function (glucocorticoids, psychotropics, narcotics, metoclopramide)
* Consumption or injection of insulin
* Apparent sensitivity to any of the study peptides as determined by the skin test

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Leslie Willis, Durham, North Carolina, United States

REFERENCES:
- [Derived] Gray SM, Hoselton AL, Krishna R, Slentz CA, D'Alessio DA. GLP-1 Receptor Blockade Reduces Stimulated Insulin Secretion in Fasted Subjects With Low Circulating GLP-1. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2500-2510. doi: 10.1210/clinem/dgac396. PMID 35775723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by advertisement from March 2017 to March 2018.
Groups:
- Sitagliptin and Non-Sitagliptin: Arms of study per sequence:
  1. Sitagliptin and Ex-9 then Saline then Non-Sitagliptin and Ex-9 then Saline 2. Sitagliptin and Saline then Ex-9 then Non-Sitagliptin and Ex-9 then Saline 3. Sitagliptin and Ex-9 then Saline then Non-Sitagliptin and Saline then Ex-9 4. Sitagliptin and Saline then Ex-9 then Non-Sitagliptin and Saline then Ex-9 5. Non-Sitagliptin and Ex-9 then Saline then Sitagliptin and Ex-9 then Saline 6. Non-Sitagliptin and Ex-9 then Saline then Sitagliptin and Saline then Ex-9 7. Non-Sitagliptin and Saline then Ex-9 then Sitagliptin and Ex-9 then Saline 8. Non-Sitagliptin and Saline then Ex-9 then Sitagliptin and Saline then Ex-9
  .
Period: Overall Study
Arm/Group | Sitagliptin and Non-Sitagliptin
Started | 40
Completed | 32
Not Completed | 8
Not completed — Failed IV access | 3
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Subjects who did not withdraw consent.
Groups:
- Sitagliptin and Non-Sitagliptin Recipients: The infusion procedures performed during study visits 2 and 3 are identical except that the oral medicine Sitagliptin will only be administered at one of the two visits, with order of Sitagliptin administration determined at random by study staff.
  Active Comparator: Sitagliptin: Subjects will receive sitagliptin prior to the start of the experiment involving 1/2 of the subjects receiving Exendin-9 (a GLP-1 receptor blocker) first over 60 minutes ; followed by a bolus arginine (5g) infusion after 30 minutes into the Ex-9 infusion, with blood draws over the next 30 minutes. Followed by a 60 minute washout and the procedure is repeated , this time with saline instead of Ex-9 (these procedures are reversed - saline first then Ex-9 - half of the time).
  Placebo Comparator - No Sitagliptin: Subjects will receive Placebo (instead of sitagliptin) prior to the start of the experiment involving 1/2 of the subjects receiving Exendin-9 (a GLP-1 receptor blocker) first over 60 minutes ; followed by a bolus arginine (5g) infusion after 30 minutes into the Ex-9 infusion, with blood draws over the next 30 minutes. Followed by a 60 minute washout and the procedure is repeated , this time with saline instead of Ex-9 (these procedures are reversed - saline first then Ex-9 - half of the time).
Arm/Group | Sitagliptin and Non-Sitagliptin Recipients
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35
Diabetes Type [Count of Participants; unit: Participants]
  No Diabetes (NDM) | 20
  Type 2 Diabetes (T2DM) | 15

OUTCOME MEASURES:

1. Primary Outcome: Arginine-stimulated Insulin Secretion With and Without GLP-1 Blockade
Description: The investigators will use the mean increment of insulin secretion rate above baseline in the 30 minutes after Arginine stimulation to integrate insulin secretion, the primary outcome measure, and 2-way ANOVA with and without Sitagliptin and Ex-9/saline at the two factors.
Time Frame: 30 minutes
Population: Participants who completed infusion protocols.
Measure: Mean (Standard Error); unit: pmol/L
Groups:
- Sitagliptin and Ex-9/Saline (Non-diabetics); Sitagliptin and Ex-9/Saline (Diabetics): The infusion procedures performed during study visits 2 and 3 are identical except that the oral medicine Sitagliptin will only be administered at one of the two visits, with order of Sitagliptin administration determined at random by study staff. In this arm, Sitagliptin will be administered.
  Active Comparator: Sitagliptin: Subjects will receive sitagliptin prior to the start of the experiment involving 1/2 of the subjects receiving Exendin-9 (a GLP-1 receptor blocker) first over 60 minutes ; followed by a bolus arginine (5g) infusion after 30 minutes into the Ex-9 infusion, with blood draws over the next 30 minutes. Followed by a 60 minute washout and the procedure is repeated , this time with saline instead of Ex-9 (these procedures are reversed - saline first then Ex-9 - half of the time).
- Non-Sitagliptin and Ex-9/Saline (Non-diabetics); Non-Sitagliptin and Ex-9/Saline (Diabetics): The infusion procedures performed during study visits 2 and 3 are identical except that the oral medicine Sitagliptin will only be administered at one of the two visits, with order of Sitagliptin administration determined at random by study staff. In this arm, placebo will be administered
  Placebo Comparator - No Sitagliptin: Subjects will receive Placebo (instead of sitagliptin) prior to the start of the experiment involving 1/2 of the subjects receiving Exendin-9 (a GLP-1 receptor blocker) first over 60 minutes ; followed by a bolus arginine (5g) infusion after 30 minutes into the Ex-9 infusion, with blood draws over the next 30 minutes. Followed by a 60 minute washout and the procedure is repeated , this time with saline instead of Ex-9 (these procedures are reversed - saline first then Ex-9 - half of the time).
Arm/Group | Sitagliptin and Ex-9/Saline (Non-diabetics) | Sitagliptin and Ex-9/Saline (Diabetics) | Non-Sitagliptin and Ex-9/Saline (Non-diabetics) | Non-Sitagliptin and Ex-9/Saline (Diabetics)
Number analyzed (Participants) | 19 | 13 | 19 | 13
pmol/L
  With GLP-1 Blockade | 320.1 (0.37) | 243.4 (0.38) | 280 (0.37) | 251.2 (0.38)
  Without GLP-1 Blockade | 318.7 (0.37) | 319.4 (0.38) | 371.4 (0.37) | 249.2 (0.38)
Statistical Analysis 1: Comparison: Sitagliptin and Ex-9/Saline (Non-diabetics) vs Non-Sitagliptin and Ex-9/Saline (Non-diabetics); Test type: Equivalence — Insulin secretion, determined by insulin or C-peptide values in the 10 minutes after arginine infusion will be compared as a repeated measure for each subject in a 2 x 2 analysis of sitagliptin/placebo and Exendin-9/saline; p < 0.05, Mixed Models Analysis; Median Difference (Final Values) = 371

ADVERSE EVENTS:
Time Frame: 1 month
Description: Presented by intervention. One subject did not receive placebo infusion.
Arm/Group | Sitagliptin | Non-Sitagliptin
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 3/35 | 2/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=35) | Non-Sitagliptin (N=34)
failed IV line (Blood and lymphatic system disorders) | 3 (3) | 2 (2) — Failure to obtain or maintain intravenous access for infusion protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT02683187/Prot_SAP_000.pdf